CLINICAL TRIAL: NCT01915719
Title: Early Non Invasive Ventilation in Immuno-compromized Patients With Acute Respiratory Failure. A Prospective Randomized Clinical Trial.
Brief Title: Early Non Invasive Ventilation in Immuno-compromized Patients With Acute Respiratory Failure.
Acronym: IVNICTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVNICTUS
Record Dates: First submitted 2013-07-26; First posted 2013-08-05 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-11

CONDITIONS: Adult; Acute Respiratory Failure Admitted in ICU; Immuno Compromized

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early non invasive ventilation (Experimental): Early non invasive ventilation
  Interventions: Procedure: Early non invasive ventilation
- Oxygen therapy only (Active Comparator): Oxygen therapy only
  Interventions: Procedure: Oxygen therapy only

INTERVENTIONS:
Procedure: Early non invasive ventilation
  Arms: Early non invasive ventilation
Procedure: Oxygen therapy only
  Arms: Oxygen therapy only

SUMMARY:
Assess the superiority of early non invasive ventilation in comparison to Oxygen therapy only, for immuno-compromized patients with acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* ICU admission
* Acute respiratory failure defined by (PaO2<60 mmHg at room air) or (polypnea >30/min or dyspnea at rest) or respiratory distress. Since less than 72 hours.
* Immuno compromized patient defined by solid tumor (treated since less than 5 years) or haematological malignancy (treated since less than 5 years) or Solid organ transplantation or Stem cell transplantation or Immunosuppressive treatment (steroid > 1mg/kg/d or >1 month or other immunosuppressive treatment >1 month)

Exclusion Criteria:

* Hypercapnia >50 mmHg or increased of hypercapnia >10 mmHg under Oxygen treatment
* Need of immediate mechanical ventilation
* Obvious cardiogenic oedema
* Vasopressor use >0.03 µg/kg/min
* Glasgow Score <13
* End of life decision
* Acute myocardial infarction
* Patient refusal
* Pregnancy
* No national health insurance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Day 28 Mortality | Day 28

SECONDARY OUTCOMES:
Needs of mechanical ventilation | Day 28
SOFA Score | Hour 72
Nosocomial infection | day 28
Length of stay in ICU | Day 28
performance status (OMS scale ranging from 0-perfect status- to 4-moribund) | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Virginie lemiale, MD, Principal Investigator — APHP
Locations (1):
- APHP, Hôpital Saint Louis, Paris, France

REFERENCES:
- [Background] Lemiale V, Resche-Rigon M, Azoulay E; Study Group for Respiratory Intensive Care in Malignancies Groupe de Recherche en Reanimation Respiratoire du patient d'Onco-Hematologie. Early non-invasive ventilation for acute respiratory failure in immunocompromised patients (IVNIctus): study protocol for a multicenter randomized controlled trial. Trials. 2014 Sep 25;15:372. doi: 10.1186/1745-6215-15-372. PMID 25257210
- [Result] Lemiale V, Mokart D, Resche-Rigon M, Pene F, Mayaux J, Faucher E, Nyunga M, Girault C, Perez P, Guitton C, Ekpe K, Kouatchet A, Theodose I, Benoit D, Canet E, Barbier F, Rabbat A, Bruneel F, Vincent F, Klouche K, Loay K, Mariotte E, Bouadma L, Moreau AS, Seguin A, Meert AP, Reignier J, Papazian L, Mehzari I, Cohen Y, Schenck M, Hamidfar R, Darmon M, Demoule A, Chevret S, Azoulay E; Groupe de Recherche en Reanimation Respiratoire du patient d'Onco-Hematologie (GRRR-OH). Effect of Noninvasive Ventilation vs Oxygen Therapy on Mortality Among Immunocompromised Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2015 Oct 27;314(16):1711-9. doi: 10.1001/jama.2015.12402. PMID 26444879